CLINICAL TRIAL: NCT01709916
Title: Comparing Diurnal Fluctuations in Intra Ocular Pressure Measured in Same Day Versus Different Days in Glaucoma Patients
Acronym: IOP
Status: Completed | Type: Observational
Sponsor: Carmel Medical Center (Other)
Responsible Party: Principal Investigator, Orna Geyer, Professor, Carmel Medical Center
Other Study IDs: CMC-11-0037-CTIL
Record Dates: First submitted 2012-10-17; First posted 2012-10-18 (Estimated); Last update posted 2015-02-24 (Estimated); Status verified 2015-02

CONDITIONS: Glaucoma
Keywords: Glaucoma; intra ocular pressure; diurnal fluctuations
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Glaucoma patients: Glaucoma patients treated with eye drops to lower the IOP.

SUMMARY:
Glaucoma is one of the leading causes of blindness in the west. The disease caused by high intra ocular pressure (IOP) and characterized by damage to the optic nerve and gradual loss of visual field. Intra ocular pressure change during the day. To evaluate the efficiency of the therapy it is common to measure the intra ocular pressure at different times of the day. Most ophthalmologists admit the patient for one day at which intra ocular pressure is measured at different times. This method does not mimic the patient daily routine and may not reflect the true diurnal fluctuations.

For this reason some ophthalmologists measure the intra ocular pressure at different times and at different days. It is not known if both methods give similar diurnal curves.

DETAILED DESCRIPTION:
A study physician will install anesthetic eye drops and will color the eye drops film with fluorescein. Study physician will use tonometer to measure the intra ocular pressure in each eye. This is a standard procedure done in any ophthalmological examination. Each patient will undergo intraocular pressure examination at 8:00, 12:00 and 16:00.

In the first day intra ocular pressure will be measured at 8:00, 12:00 and 16:00, same day measurements. The day after intra ocular pressure will be measured at 8:00, two days after at 12:00 and three days after at 16:00. One month later the patient will undergo another serious of intra ocular pressure measurements.

In the first day intra ocular pressure will be measured at 8:00, 12:00 and 16:00, same day measurements. The day after intra ocular pressure will be measured at 8:00, two days after at 12:00 and three days after at 16:00.

The relationship between the two diurnal curves will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Glaucoma patient.
* Age 18-80 years
* Able to read and understand Hebrew, able to sign informed consent in Hebrew.

Exclusion Criteria:

* Ophthalmic laser treatment or surgery 3 months prior to enrollment.
* Eye infection or inflammation.
* Corneal pathology altering IOP measurement.
* Patients not cooperating during IOP measurement.
* non compliant patients

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Glaucoma patients using eye drops to lower intra ocular pressure.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2012-11; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
IOP at different times of the day at same day versus different times and different days | 5 weeks
  measurements of intra ocular pressure at different times of the day at same day versus different times and different days.

CONTACTS AND LOCATIONS:
Overall Officials: Orna Geyer, MD, Principal Investigator — Carmel Medical Center
Locations (1):
- Carmel Medical Center, Haifa, Israel